CLINICAL TRIAL: NCT04604106
Title: General Anesthesia Exposure and Neurodevelopmental Outcome in Pediatrics
Acronym: GAP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Sanne Maat, Dr. J.P.M. Derikx, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL71873.018.19
Record Dates: First submitted 2020-10-21; First posted 2020-10-27 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Anesthesia; Infant Development; Anesthesia; Adverse Effect
Keywords: Anesthesiology; Neuropsychological test; Infant neurodevelopmental disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient group: Infant aged 12 months (± four weeks) with a history of general anesthesia exposure
  Interventions: Diagnostic Test: Eyetracker; Diagnostic Test: Ages & Stages questionnaire; Diagnostic Test: Bayley Scale of Infant Development
- Healthy subject group: Infant aged 12 months (± four weeks) without a history of general anesthesia
  Interventions: Diagnostic Test: Eyetracker; Diagnostic Test: Ages & Stages questionnaire; Diagnostic Test: Bayley Scale of Infant Development

INTERVENTIONS:
Diagnostic Test: Eyetracker — Eye-tracking is an objective, non-invasive method and particularly suited to assess neurodevelopmental outcome in infants.
Diagnostic Test: Ages & Stages questionnaire — The Ages & Stages Questionnaire is a conventional instrument used to measure developmental outcome in infants.
Diagnostic Test: Bayley Scale of Infant Development — The Bayley Scale of Infant Development is a conventional instrument used to measure developmental outcome in infants.

SUMMARY:
This study investigates the impact of different levels of anesthesia exposure on children's neurocognitive development and evaluates the concurrent validity of different methods that assess neurodevelopmental outcome.

DETAILED DESCRIPTION:
The US Food and Drug Administration (FDA) recently released an official warning regarding the potentially harmful impact of repeated and prolonged (more than three hours) general anesthesia on the child's brain. The potential impact of anesthesia highlights the importance of remediating the need for repeated and prolonged surgery with accompanying anesthesia exposure in a time of cerebral vulnerability and if possible, delay exposure to avoid potentially preventable harm. Therefore, it is crucial to better understand the impact of (different durations and frequencies of) anesthesia exposure on neurodevelopment.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 months (± four weeks) with a history of general anesthesia exposure (patient group) or without a history of general anesthesia (healthy controls)

Exclusion Criteria:

* Children with comorbid conditions affecting structure and/or function of the central nervous system (e.g. premature birth) will be excluded from participation in this study.

Ages: 11 Months to 13 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: At the outpatient clinic of the department of pediatric surgery, children (< 12 months old) who are scheduled for or already underwent a single short, long or repetitive general anesthesia will be identified by the (fellow) pediatric surgeon. Parents/caretakers will be asked to participate in this study by the (fellow) surgeon who will ask informed consent. Healthy controls exist of eligible acquaintances and children that will be recruited via child health care centres by a member of the research team
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2020-10-21 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive development as measured using eye-tracking metrics | At the age of 12 months (± four weeks)
  Neurocognitive development as measured using eye-tracking metrics

SECONDARY OUTCOMES:
Conventional measures of neurocognitive development (Ages & Stages Questionnaire and Bayley Scales of Infant Development ) | At the age of 12 months (± four weeks)
  Neurocognitive development as measured using the Ages & Stages Questionnaire and Bayley Scales of Infant Development
Total anesthesia time. | At the age of 12 months (± four weeks)
  Surgery and anesthesia time will be recorded by the (fellow) surgeon performing the operation(s). When multiple procedures are carried out, durations will be combined and these results will be retrieved during analysis of the data.

CONTACTS AND LOCATIONS:
Overall Officials: J.P.M. Derikx, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); J. Oosterlaan, Prof., Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Amsterdam UMC, locatie AMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes